CLINICAL TRIAL: NCT06703528
Title: Cryoablation System with Liquid Nitrogen for the Treatment of Atrial Fibrillation
Brief Title: An Exploratory Clinical Study to Evaluate the Safety and Efficacy of a Cardiac Surgical Cryoablation System for the Treatment of Atrial Fibrillation
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-2413
Record Dates: First submitted 2024-11-16; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (AF); Heart Valve Diseases
Keywords: atrial fibrillation; heart valve diseases
MeSH Terms: conditions — Atrial Fibrillation; Heart Valve Diseases | interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: cryoablation — The therapeutic cryoablation agent used in this trial was liquid nitrogen with an evaporation temperature of -196°C, which was transported to the ablation pen through a vacuum line to exchange energy at the heart site to perform cryoablation.

SUMMARY:
The goal of this prospective, observational study is to evaluate the safety and efficacy of a cardiac surgical cryoablation system for the treatment of atrial fibrillation. This study will be conducted at Fuwai Hospital in China. A total of 10 subjects with heart valve diseases (e.g., mitral, tricuspid, and aortic valve diseases) requiring surgical treatment and with atrial fibrillation will be enrolled in the study, and all of them will undergo surgical ablation using surgical cryoablation devices (cryoablation clamps and pens) with follow-up visits at 3 and 6 months after the procedure. In this study, the incidence of cardiac and cerebrovascular-related adverse events in the perioperative period and at 6 months after procedure is defined as the primary safety endpoint (all-cause mortality, stroke, systematic embolism, cardiac reoperations, heart failure requiring hospitalization, ablation-related coronary artery stenosis/occlusion, pulmonary vein stenosis, and rate of permanent pacemaker implantation.). The primary efficacy endpoint is the probability of freedom from atrial tachyarrhythmias at 6 months after the procedure. Device ease of use, technical success, ablation procedure time, and assessment of the incidence of device defects are defined as secondary endpoints.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most important causes of ischemic stroke, which is a serious danger to human health. Heart valve disease, especially mitral valve lesions, often secondary to AF, thrombus formation in the cardiac cavity, embolus dislodgement can lead to embolic complications. Some studies have reported that in mitral valve surgery 40%-60% of patients can be combined with AF. For the treatment of AF, Cox maze III has become the standard surgical procedure for the treatment of AF due to its excellent efficacy. However, due to the complexity of surgical operation and many postoperative complications, it has not been widely promoted.Cox maze IV surgery is based on the Cox maze III procedure, which utilizes a new energy source instead of the traditional "cut and sew" to form a specific ablation line in the atria to eliminate AF and restore the sinus rhythm, which is easy to operate and can achieve the same results as the Cox maze III procedure. It is widely accepted because it is easy to operate and can achieve similar clinical efficacy as Cox maze III.

Currently widely used in clinical treatment of Cox maze IV procedure is mostly completed by radiofrequency combined with cryoablation or cryoablation alone. Cryoablation has different thermal effects compared with radiofrequency ablation, and the cells within the ablation line undergo apoptosis, but the cell structure is preserved, which is not easy to cause coronary stenosis or spasm; it is not limited by the incision, and all the ablation lines can be completed in the cardiac cavity, which overcomes the limitations of the minimally invasive surgery for the exposure of the left posterior wall of the left atrium.

Currently on the market are Medtronic's Cardioblate CryoFlex and AtriCure's CryoICE, both of which utilize the principle of high-pressure gas throttling and refrigeration to achieve cryoablation.The Cardioblate CryoFlex utilizes high-pressure argon gas at 310-410 atmospheres, with a minimum temperature of -150°C. CryoICE utilizes high-pressure nitrous oxide at 69 atmospheres, with a minimum temperature of -70°C. Due to the relatively high treatment temperature of these two products, the wall penetration time is longer and the maximum ablation depth is smaller, which can easily lead to incomplete ablation. At the same time, high-pressure gas is likely to cause equipment operation safety risks, work noise is larger. Nitrous oxide, as a kind of anesthesia gas with toxic effect on human body, has poor environmental friendliness, cannot be discharged arbitrarily.

The therapeutic agent used in the cryoablation in this study is liquid nitrogen with an evaporation temperature of -196°C. It is transported to the ablation clamp and pen through a vacuum pipeline to carry out energy exchange in the cardiac area and implement cryoablation. According to the test results, the cooling speed of this product is about 30s, and the temperature distribution of the ablation clamp and pen in the treatment area is uniform, with a difference of no more than 5℃, which can realize convenient, fast and effective ablation. At the same time, the price of liquid nitrogen is cheap and easy to obtain, which is easy to be promoted in large, medium and small cities across the world, benefiting the majority of patients with AF.

In the previous period, the investigators have applied cryoablation clamps and ablation pens for animal experiments, and the results have reached the expectation. However, it is not yet clear whether this cryoablation device can obtain better safety and efficacy in AF patients. Therefore, the present study is intended to evaluate the safety and efficacy of the cardiac surgical cryoablation device through a small sample size single-arm exploratory clinical trial, so as to lay the foundation for the subsequent widespread clinical application of this cryoablation device.

ELIGIBILITY:
Inclusion Criteria:

* patients with valvular disease (e.g., mitral, tricuspid, and aortic valve disease) requiring surgical intervention;
* patients with atrial fibrillation who consent to cryoablation;
* 18-75 years of age (as of the date of signing the informed consent form);
* signing the patient's informed consent.

Exclusion Criteria:

* intracardiac thrombosis;
* patients with absolute contraindications to anticoagulation;
* combination of other cardiac diseases requiring surgical treatment;
* patients with a diagnosis of coronary artery disease (coronary artery enhancement CT or coronary angiography suggesting that any one of the three coronary vessels and their major branches has a stenosis greater than or equal to 50%);
* patients with generalized malignant disease or severe insufficiency of liver, kidney, heart and lung functions;
* patients with current active infection;
* pregnant and lactating patients;
* patients with a prior history of cardiac surgery;
* patients with myocardial infarction within the last 3 months;
* patients who have suffered a stroke within the last 3 months;
* patients with an anterior-posterior left atrial diameter greater than 70 mm;
* left ventricular ejection fraction (LVEF) <50%;
* patients who are not expected to complete the 6-month postoperative follow-up;
* those who are participating in other clinical trials and have not met the primary endpoint;
* those who, in the opinion of the investigator, are not suitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are aged between 18-75 years old, with heart valve disease requiring surgery and combined with atrial fibrillation, no previous cardiac surgery, no myocardial infarction or stroke within 3 months, no absolute contraindications to anticoagulation, no other cardiac disease that does not require surgical treatment, no diagnosis of coronary artery disease, no active infections, no serious insufficiency of the liver, kidneys, cardiopulmonary function, no thrombus in the cardiac cavity, and the internal diameter of left atrium is no more than 70mm and the left ventricular ejection fraction is not less than 50%.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Perioperative and 6-month postoperative cardiac and cerebrovascular-related adverse event rates | From enrollment to the end of the trial at 6 months
  Cardiac and cerebrovascular-related adverse events included all-cause mortality, stroke, systematic embolism, repeat cardiac surgery, heart failure requiring hospitalization, ablation-related coronary artery stenosis/occlusion, pulmonary vein stenosis, and permanent pacemaker implantation rates.
The probability of freedom from atrial tachyarrhythmias at 6 months after cryoablation | From enrollment to the end of the trial at 6 months
  The probability of freedom from atrial fibrillation, atrial flutter, and atrial tachycardia in the absence of class I/III antiarrhythmic drugs at 6 months postoperatively.

IPD SHARING:
Plan to Share IPD: No